CLINICAL TRIAL: NCT05530421
Title: Selinexor, Venetoclax, and Dexamethasone (XVenD) in t(11;14)-Positive Relapsed/Refractory Multiple Myeloma (SELVEDge Study)
Brief Title: Selinexor, Venetoclax, and Dexamethasone (XVenD) in t(11;14)-Positive Relapsed/Refractory Multiple Myeloma
Acronym: SELVEDge
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Dickran Kazandjian, MD, Professor of Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220595
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — selinexor; venetoclax; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- XVenD Group (Experimental): Participants will receive XVenD combination therapy of Selinexor (X), Venetoclax (Ven) and Dexamethasone (D) orally during each 28-day cycle. Doses will be administered as follows:
  * Cycle 1 Days 1 to 7:
    * Venetoclax 400 mg orally (PO), Days 1-7
    * Dexamethasone 40 mg PO, Day 1
  * Cycle 1 Days 8 to 28:
    * Venetoclax 800 mg PO, Days 8-28
    * Dexamethasone 40 mg PO, Days 8, 15, and 22
  * Cycles 2 to 4:
    * Selinexor 80 mg PO, Days 1, 8, 15, and 22
    * Venetoclax 800 mg PO, Days 1-28
    * Dexamethasone 40 mg PO, Days 1, 8, 15, and 22
  * Cycle 5 and beyond:
    * Selinexor 80 mg PO, Days 1, 8, 15, and 22
    * Venetoclax 800 mg PO, Days 1-28
    * Dexamethasone 20 mg PO, Days 1, 8, 15, and 22
  Selinexor dose will be reduced to 60 mg for remaining participants if after the first 6 participants complete the first cycle and 2 or more out of these first 6 participants experience dose-limiting toxicities (DLTs).
  Interventions: Drug: Selinexor; Drug: Venetoclax; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor tablets will be administered orally (PO) once per day at assigned dosage and frequency per protocol.
  Other Names: Xpovio
Drug: Venetoclax — Venetoclax tablets will be administered orally (PO) once per day at assigned dosage and frequency per protocol.
  Other Names: Venclexta; Venclyxto
Drug: Dexamethasone — Dexamethasone tablets will be administered orally (PO) once per day at assigned dosage and frequency per protocol.
  Other Names: Decadron; Ozurdex; Dexycu

SUMMARY:
The purpose of this research is to determine whether the combination of selinexor, venetoclax, and dexamethasone therapy can increase anti-cancer effects in patients with translocation 11;14-positive (t(11;14)), relapsed/refractory myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a documented diagnosis of multiple myeloma defined by the International Myeloma Working Group Criteria (IMWG).5 Patients at initial diagnosis must have had a serum M-protein ≥ 3 g/dL and/or bone marrow plasma cells ≥10%, and at least one of the following:

   1. Anemia: Hemoglobin ≤10 g/dL, or
   2. Renal failure: serum creatinine ≥ 2.0 mg/dL, or
   3. Hypercalcemia: Ca ≥10.5 mg/dL, or
   4. Lytic bone lesions on X-ray, CT, or Positron emission tomography/Computed Tomography (PET/CT), or
   5. ≥ 2 focal lesions on spinal magnetic resonance imaging (MRI), or
   6. ≥ 60% bone marrow plasma cells, or Involved/un-involved serum free light chain ratio ≥ 100. Age ≥18 years of age on day of signing informed consent.
2. Patients must have had a bone marrow (BM) biopsy proven plasma cell myeloma harboring the t(11;14) translocation as reported by a Clinical Laboratory Improvement Amendments (CLIA) certified assay (i.e. local fluorescence in situ hybridization (FISH) testing). BM biopsy can be performed at time of enrollment or documented FISH results (i.e. original FISH report) can be used.
3. Must have Relapsed or Relapsed and Refractory Multiple Myeloma. Patients must have documented evidence of having received two prior lines of therapy and be refractory to, not a candidate for (ineligible), or intolerant of at least one immunomodulatory (IMiD), one proteasome inhibitor, and one anti-cluster of differentiation 38 (anti-CD38) monoclonal antibody-based treatments.
4. Documented measurable disease based on the IMWG guidelines within the 4 weeks prior to registration defined by any one of the following criteria:

   1. Serum monoclonal protein ≥ 0.5 g/dl
   2. Urine monoclonal protein >200 mg/24 hour
   3. Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio
   4. Bone marrow plasma cells ≥ 30%
   5. A measurable lesion on PET/CT or MRI ≥ 2 cm
5. Be ≥ 18 years of age on day of signing informed consent
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of ≤ 3 (Appendix A)
7. Adequate organ function as evidenced by the following laboratory parameters within 4 weeks of C1D1:

   Hematologic:
   1. Absolute neutrophil count (ANC) 1000/microliter (mcL) (granulocyte-colony stimulating factor (G-CSF) allowed)
   2. Platelets ≥ 50,000/mcL (transfusions and stimulators permitted); in patients with >50% bone marrow plasma cells, platelets ≥ 30,000/mcL
   3. Hemoglobin ≥ 8 g/dL (transfusions permitted)

      Non-hematologic:
   4. Serum creatinine ≤ 1.5 X ULN (except if due to myeloma) or calculated creatinine clearance (CrCl)/Estimated glomerular filtration rate (eGFR) (by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI), Modification of Diet in Renal Disease (MDRD), or Cockcroft-Gault) ≥ 15 mL/min/1.73 m2
   5. Serum total bilirubin ≤ 1.5 X ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 X ULN)
   6. Aspartate transaminase (SGOT) and alanine transaminase (SGPT) ≤ 2.5 X ULN
8. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 90 days following the last dose of study treatment.
9. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.

Exclusion Criteria:

1. Has received selinexor or another specific inhibitor of nuclear exporter (SINE) compound previously.
2. Has any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
3. Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to Cycle 1 Day 1 (C1D1). Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to C1D1 are acceptable.
4. Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
5. Pregnant or breastfeeding females.
6. Active, unstable cardiovascular function, as indicated by the presence of symptomatic ischemia, or Uncontrolled clinically significant conduction abnormalities (eg, patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or Congestive heart failure of New York Heart Association Class ≥3 or known left ventricular ejection fraction <40%, or Myocardial infarction within 3 months prior to C1D1.
7. Subjects with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for >8 weeks and viral load is <100 IU/ml prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed. Subjects with Human Immunodeficiency Virus (HIV) who have cluster of differentiation 4-positive (CD4+) T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections in the last year are allowed.
8. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
9. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Comprehensive Cancer Network® (NCCN) Clinical Practice Guidelines in Oncology (CPGO) (https://www.nccn.org/guidelines/category_3) for antiemesis and anorexia/cachexia (palliative care).
10. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
11. Contraindication to any of the required concomitant drugs or supportive treatments.
12. Patients unwilling or unable to comply with the protocol or known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-03-26 (Estimated)

PRIMARY OUTCOMES:
Fraction of Participants Achieving Overall Response | Up to 3 years
  Overall response rate (ORR) will be reported as the fraction of participants achieving either complete response (CR) or partial response (ORR = CR + PR) to study treatment. Response to therapy will be assessed by treating physician using International Myeloma Working Group 2016 response criteria.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 3 years
  Duration of response is defined as the elapsed time from date of partial response (PR) or better to the date of progressive disease (PD) or death, whichever is first.
Minimal Residual Disease Negative Complete Response Rate | Up to 3 years
  Minimum residual disease negative (MRD negative) complete response (CR) rate will be reported as the fraction of participants achieving CR who show less than one myeloma cell per million bone marrow cells after protocol therapy. Response to therapy will be assessed using International Myeloma Working Group 2016 response criteria.
Progression-Free Survival (PFS) | Up to 3 years
  Progression-free survival (PFS) will be defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first. For surviving participants without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) will be defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact.
Rate of Treatment-Emergent Adverse Events | Up to 10 months
  Safety and tolerability of assigned protocol treatment will be reported as the rate of treatment-related toxicity, including serious adverse events (SAEs), grade 3 or higher adverse events, and all-grade adverse events (AEs), in study participants using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, as assessed by treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Dickran Kazandjian, MD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - University of Miami, Lennar Foundation Medical Center, Coral Gables, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami, Sylvester Comprehensive Cancer Center, Miami, Florida

IPD SHARING:
Plan to Share IPD: No